CLINICAL TRIAL: NCT00510562
Title: Effect of Cranial Osteopathy on Visual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Mark Sandhouse, Associate Professor & Chair, Department of OPP, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPD-COM 06200101
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Visual Function
Keywords: Cranial manipulation; Visual function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Assessment for cranial strain patterns, followed by indirect osteopathic treatment of dysfunctions found on assessment, followed by reassessment.
  Interventions: Procedure: Cranial osteopathic manipulation
- 2 (Sham Comparator): Assessment for cranial strain patterns, followed by laying on of hands, followed by reassessment.
  Interventions: Procedure: Sham/Placebo

INTERVENTIONS:
Procedure: Cranial osteopathic manipulation — This treatment is performed by exaggerating the motion asymmetry with a minimum of pressure (a few ounces) and holding the position until the motion becomes symmetrical.
  Arms: 1
Procedure: Sham/Placebo — A laying on of hands with no treatment being performed.
  Arms: 2

SUMMARY:
It is the purpose of this study to attempt to determine if there is an immediate, measurable change in visual function as a direct result following a session of cranial osteopathic manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Free of active ocular or systemic disease
* Refractive error between six diopters of myopia and five diopters of hyperopia with regular astigmatism of any amount
* Normal best-corrected visual acuity at 20/40 or better
* Normal amplitude of accommodation
* Willing to undergo cranial osteopathic manipulation

Exclusion Criteria:

* Pregnancy
* History of previous closed head trauma or brain injury
* Students from the Nova Southeastern University Colleges of Osteopathic Medicine and Optometry
* Prior cranial manipulative treatment/craniosacral therapy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2001-10; Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Accommodative system testing Visual acuity testing Stereoacuity testing Vergence system testing Pupillary testing | Immediately after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sandhouse, D.O., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University Davie Health Center, Fort Lauderdale, Florida, United States

REFERENCES:
- [Derived] Sandhouse ME, Shechtman D, Sorkin R, Drowos JL, Caban-Martinez AJ 3rd, Patterson MM, Shallo-Hoffmann J, Hardigan P, Snyder A. Effect of osteopathy in the cranial field on visual function--a pilot study. J Am Osteopath Assoc. 2010 Apr;110(4):239-43. PMID 20430912